CLINICAL TRIAL: NCT04509804
Title: Target Gene Sequencing for Advanced Stage, Relapsed/Refractory Natural Killer/T-cell Lymphoma and the Correlation Between Gene Abmormalities and Chemotherapy Efficacy
Brief Title: Target Gene Sequencing for Advanced Stage, Relapsed or Refractory Natural Killer/T-cell Lymphoma
Status: Completed | Type: Observational
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mei Dong, Principal Investigator, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: GeneNKT
Record Dates: First submitted 2018-08-07; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Lymphoid Neoplasm

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non-interventional — non-interventional

SUMMARY:
Although modern radiation techniques combined with chemotherapy has greatly improved the local control and long-term survivals for patients with early-stage NKTCL, relapse and systemic dissemination are common for localized patients. Relapsed/refractory diseases together with advanced stage NKTCLs uaually progress rapidly with poor prognosis (5-year overall survival rate, 0-20%). According to published studies, some recurrent genetic alternations have been identified in NKTCL, including oncogene/tumor suppressive gene abberants, epigenetic changes, cellular signaling pathways abnormalities, cellular apoptosis related genes and so forth. However, the gene profiling techniques and materials vary in different studies, no consensus has been reached on the gene abnormalities of advanced, or relapsed/refractory NKTCL up to now. Additionally, gene sequencing using ctDNA of peripheral blood has been unexploited in NKTCL patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of NKTCL with typical morphology and immunophenotype, according to the 2008 World Health Organization classification of lymphomas;
2. stage III/IV disease; or relapsed or refractory disease after at least one line prior teratment;
3. age ≥ 18 years;
4. ECOG performance status 0-2;
5. at least one measurable lesion;
6. adequate hematological, hepatic, and renal functions;
7. life expectancy of more than 3 months.

Exclusion Criteria:

1. Previously untreated stage I/II disease;
2. with no adequate tumour tissue;
3. any coexisting medical problems of sufficient severity to prevent full compliance with the study protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We plan to recurit 30 eligile patients who are diagnosed in our hospital.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Concordance | 2 years
  The concordance of plasma cfDNA genotyping and tumor genotyping is defined as the ratio of gene variants detected in tumor and cfDNA to variants identified in tumor

CONTACTS AND LOCATIONS:
Locations (1):
- Mei Dong, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided